CLINICAL TRIAL: NCT01640379
Title: Technology Enhanced Community Health Nursing (TECH-N) to Prevent Recurrent Sexually Transmitted Infections After Pelvic Inflammatory Disease
Brief Title: Technology Enhanced Community Health Nursing (TECH-N) Study
Acronym: TECH-N
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NA_00068846; 1R01NR013507-01 (NIH)
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Pelvic Inflammatory Disease (PID)
Keywords: Pelvic Inflammatory Disease (PID); Community Health Nursing; Text Messaging; mobile health (mhealth); Adolescents
MeSH Terms: conditions — Pelvic Inflammatory Disease | interventions — Spermine Synthase

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TECH-N (Experimental): Participants receive the Technology Enhanced Community Health Nursing Visit (CHN) within 5 days during which Sister to Sister and clinical assessment performed and text-messaging support
  Interventions: Behavioral: Technology Enhanced Community Health Nursing
- Control (No Intervention): Participants receive enhanced standard of care

INTERVENTIONS:
Behavioral: Technology Enhanced Community Health Nursing — * Text-messaging (twice daily medication reminders w/ positive adherence messages, positive sexual health messages throughout the 30 day treatment period)
  * Enhanced community health nursing visit on day 3-5, includes evidence-based STI/HIV prevention component (Sister to Sister Teen)
  Other Names: Sister to Sister Teen; Short Messaging System (SMS) communication (Text Messages)
  Arms: TECH-N

SUMMARY:
The investigators are enrolling 350 young women 13-25 years old diagnosed with pelvic inflammatory disease (PID) in Baltimore and randomize them to receive community health nurse (CHN) clinical support using a single post-PID face-to-face clinical evaluation and short messaging system communication support during the 30. The investigators hypothesize that repackaging the recommended Centers for Disease Control and Prevention (CDC) follow-up visit using a technology-enhanced community health nursing intervention (TECH-N) with integration of an evidence-based sexually transmitted infection (STI) prevention curriculum will reduce rates of short-term repeat infection by improving adherence to PID treatment and reducing unprotected intercourse and be more cost-effective compared with outpatient standard of care (and hospitalization).

DETAILED DESCRIPTION:
Pelvic Inflammatory Disease (PID) remains a serious reproductive health disorder and disease rates remain unacceptably high among minority adolescent girls and young adult women. Each episode of this upper reproductive tract infection, usually caused by a sexually transmitted infection (STI), increases the risk for multiple sequelae including tubal infertility, ectopic pregnancy, and chronic pelvic pain (CPP). Previous research demonstrates that inpatient treatment for PID is expensive without incremental increases in effectiveness when compared with outpatient treatment. The investigators' work and that of others suggest that additional outpatient cost-effective PID health care supports are needed for this vulnerable population to improve short and long-term reproductive health outcomes, including recurrent sexually transmitted infection and PID.

Prior research has also demonstrated that community health nurse (CHN) interventions can increase access to appropriate resources enhance health care utilization and promote risk-reducing behavior. The investigators propose that integrating a technology component conducted by the CHN will increase appeal to adolescent females. The investigators' pilot data of a text messaging intervention for reproductive health clinical reminders has demonstrated that use of cell phones to assist urban adolescents residing in high STI prevalent communities with self-care is both highly acceptable and feasible.

The investigators hypothesize that repackaging the recommended CDC-follow-up visit using a technology-enhanced community health nursing intervention (TECH-N) with integration of an evidence-based STI prevention curriculum will reduce rates of short-term repeat infection by improving adherence to PID treatment and reducing unprotected intercourse and be more cost-effective compared with outpatient standard of care (and hospitalization). We are enrolling 350 young women 13-21years old diagnosed with PID in Baltimore and randomizing them to receive CHN clinical support using a single post-PID face-to-face clinical evaluation and SMS communication support during the 30-days following the PID diagnosis or optimized standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Mild-moderate PID
* Outpatient treatment disposition
* Permanently reside in the Baltimore Metropolitan area
* Willing to sign informed consent & be randomized

Exclusion Criteria:

* Pregnant
* Concurrent diagnosis of Sexual Assault
* Unable to communicate/complete study procedures

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 286 (Actual)
Dates: Start 2012-07; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Trent, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Trent M, Yusuf HE, Perin J, Anders J, Chung SE, Tabacco-Saeed L, Rowell J, Huettner S, Rothman R, Butz A, Gaydos CA. Clearance of Mycoplasma genitalium and Trichomonas vaginalis Among Adolescents and Young Adults With Pelvic Inflammatory Disease: Results From the Tech-N Study. Sex Transm Dis. 2020 Nov;47(11):e47-e50. doi: 10.1097/OLQ.0000000000001221. PMID 32569258
- [Derived] Trent M, Perin J, Gaydos CA, Anders J, Chung SE, Tabacco Saeed L, Rowell J, Huettner S, Rothman R, Butz A. Efficacy of a Technology-Enhanced Community Health Nursing Intervention vs Standard of Care for Female Adolescents and Young Adults With Pelvic Inflammatory Disease: A Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e198652. doi: 10.1001/jamanetworkopen.2019.8652. PMID 31390037
- [Derived] Ha MM, Belcher HME, Butz AM, Perin J, Matson PA, Trent M. Partner Notification, Treatment, and Subsequent Condom Use After Pelvic Inflammatory Disease: Implications for Dyadic Intervention With Urban Youth. Clin Pediatr (Phila). 2019 Oct;58(11-12):1271-1276. doi: 10.1177/0009922819852979. Epub 2019 Jun 5. PMID 31165630
- See also: JHU Institute for Clinical and Translational Research (ICTR) Registry Link — http://trials.johnshopkins.edu/studyData.cfm?sdUUID=5C9058B4-AB34-F039-B91E08D4E7B76258

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Experimental: TECH-N Participants receive the Technology Enhanced Community Health Nursing Visit (community health nursing visits within 5 days during which Sister to Sister and clinical assessment performed and text-messaging support
Period: Overall Study
Arm/Group | Intervention | Control
Started | 149 | 137
Completed | 135 | 125
Not Completed | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 149 | 137 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.6 (2.4) | 18.8 (2.4) | 18.7 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 137 | 286
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 136 | 126 | 262
  White | 3 | 2 | 5
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 149 | 137 | 286
Positive Sexually Transmitted Infection Test (GC or CT) [Count of Participants; unit: Participants] — Positive sexually transmitted infection test for gonorrhea (GC) or chlamydia (CT) Population: Some baseline tests are inconclusive because the sample was not usable, so only 269 out of 286 have results.
  Participants
    number analyzed (Participants) | 142 | 127 | 269
    (all) | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Sexually Transmitted Infection Test (STI)
Description: STI testing (positive Neisseria gonorrhoeae (GC) or Chlamydia trachomatis CT) tested at 90 days using nucleic acid amplification testing (NAAT).
Time Frame: 90 Days
Population: Adolescent and young adult women with pelvic inflammatory disease (PID) in Baltimore City randomized to the intervention or control group and also had results for chlamydia (CT) and gonorrhea (GC) at 90 days after enrollment. All enrolled participants were followed as long as possible for entire 90 days.
Measure: Count of Participants; unit: Participants
Groups:
- TECH-N: Participants receive the Technology Enhanced Community Health Nursing Visit (community health nursing visits within 5 days during which Sister to Sister and clinical assessment performed and text-messaging support
  Technology Enhanced Community Health Nursing: -Text-messaging (twice daily medication reminders w/ positive adherence messages, positive sexual health messages throughout the 30 day treatment period)
  -Enhanced community health nursing visit on day 3-5, includes DEBI STI/HIV prevention component (Sister to Sister Teen)
Arm/Group | TECH-N | Control
Number analyzed (Participants) | 135 | 125
Participants | 6 | 13
Statistical Analysis 1: Comparison: TECH-N vs Control; A comparison of Chlamydia or Gonorrhea positivity at 90 days post intervention; Test type: Superiority; p = 0.070, t-test, 2 sided — Judged by type one error limit alpha = 0.05; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.15 to 1.09] — The odds ratio is for the difference in chlamydia or gonorrhea (CT/GC) rates between arms at ninety days after intervention
Statistical Analysis 2: Comparison: TECH-N vs Control; We used generalized estimating equations to test for a difference in the trend of chlamydia or gonorrhea (CT/GC) rates over the study period. The null hypothesis is that rates of CT/GC for women in the intervention arm were changing over the study period similarly to CT/GC rates in the control arm; Test type: Superiority; p = 0.043, generalized estimating equations — Judged by type one error limit alpha = 0.05; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.39 to 0.98] — The odds ratio is for the difference in rate of change over time between arms, so is the difference in the odds increment for those receiving TECH N intervention versus the control group

2. Secondary Outcome: Number of Participants That Adhered to Self-treatment
Description: Completion of 72-hour assessment visit by medical provider, medication adherence (self-reported), partner notification, partner treatment, and temporary sexual abstinence
Time Frame: Day 15
Population: Chi-square test results from participants in the intervention and control groups who had data on adherence to treatment. Out of 149 enrolled in the intervention arm, 10 were lost to followup by 72 hours. Out of 137 enrolled in the control arm, 15 were lost by 72 hours and so are missing this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- TECH-N: Participants receive the Technology Enhanced Community Health Nursing Visit (community health nursing visits within 5 days during which Sister to Sister and clinical assessment performed and text-messaging support
  Technology Enhanced Community Health Nursing: -Text-messaging (twice daily medication reminders w/ positive adherence messages, positive sexual health messages throughout the 30 day treatment period)
  -Enhanced community health nursing visit on day 3-5, includes evidence-based STI/HIV prevention component (Sister to Sister Teen)
Arm/Group | TECH-N | Control
Number analyzed (Participants) | 139 | 123
Participants | 131 | 20
Statistical Analysis 1: Comparison: TECH-N vs Control; H0: Women in TECHN arm had 72 hour visit with same frequency as women in control arm; Test type: Superiority; p < 0.001, Chi-squared; Adjusted for age, debut age, number of lifetime partners, baseline STI status (any vs none), insurance, and if woman had prior pregnancy; Odds Ratio (OR) = 92.2, 95% CI 2-sided [37.0 to 230.1] — Odds ratio is interpretable as the expected chance of having a 72 follow-up for intervention women compared to women in the control arm, given similar age, debut age, number of lifetime partners, baseline STI status, insurance, and pregnancy history
Statistical Analysis 2: Comparison: TECH-N vs Control; H0: Women in TECHN arm reported complete adherence to medication regimen (yes or no) with same frequency as women in control arm; Test type: Superiority; p = 0.084, Regression, Logistic; Adjusted for age, debut age, number of lifetime partners, pregnancy history, baseline STI status (any versus none), and insurance; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.36 to 1.05] — Odds ratio is for intervention arm relative to control
Statistical Analysis 3: Comparison: TECH-N vs Control; H0: Women in TECHN arm notified their partners about their diagnoses more often than women in the control arm; Test type: Superiority; p = 0.867, Regression, Logistic; [statistical method as in outcome 2, analysis 2]; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.36 to 2.34] — Odds ratio is for the chances of partner notification among TECH N recipients, relative to those in control arm
Statistical Analysis 4: Comparison: TECH-N vs Control; H0: Partners of women receiving the TECH-N intervention were treated more often than the partners of women in the control arm; Test type: Superiority; p = 0.153, Regression, Logistic; [statistical method as in outcome 2, analysis 2]; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.33 to 1.19] — Odds ratio is for partners of TECH-N recipients versus partners of women in control arm
Statistical Analysis 5: Comparison: TECH-N vs Control; H0: Women in the TECHN arm practiced temporary sexual abstinence for two weeks after their diagnosis more often than those in the control arm; Test type: Superiority; p = 0.351, Regression, Logistic; [statistical method as in outcome 2, analysis 2]; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.86 to 1.06] — Odds ratio is for women in the TECH-N arm relative to women in the control arm

ADVERSE EVENTS:
Time Frame: Women were followed for adverse events for the primary study period of three months.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/137
Other Adverse Events (participants affected / at risk) | 1/149 | 0/137
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=149) | Control (N=137)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Enrolled participant diagnosed with pregnancy after enrollment, and positive for sexually transmitted infection. The patient could not be reached after multiple attempts and certified letters sent to patient and primary care provider (PCP).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT01640379/Prot_SAP_000.pdf